CLINICAL TRIAL: NCT02118051
Title: Prospective Randomized Study for the Evaluation of Controlled Ovarian Stimulation With Corifollitropin Alpha in Patients With Expected or Poor Ovarian Response in IVF Cycles
Brief Title: Effect of Treatment With Corifollitropin Alpha in Vitro Fertilization in Patients With Poor Ovarian Response.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POR-ELONVA; 2013-002027-42 (EudraCT Number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2016-09

CONDITIONS: Infertility
Keywords: Infertility; IVF; Corifollitropin Alfa treatment; Ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — ganirelix; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CFA , hMG,Ganirelix,choriogonadotropin alfa,progesterone. (Experimental): Corifollitropin Alfa (CFA) 150 ug from the 2nd day of the cycle for 7 days. hMG 300 IU/24h, if required from the 8th day of the Controlled Ovarian Stimulation , until the day human chorionic gonadotropin ( hCG.) Ganirelix 0.25 mg,Dose: 250μg/24h since the day observe a follicle> 14mm. Recombinant choriogonadotropin alfa,Dose: 6,500 IU, pods, when follicles> 17 mm are observed.
  Micronized natural progesterone. Route of administration: vaginal. Dose: 400mg/24, from embryo transfer until the day of b-hCG.
  Interventions: Drug: Ganirelix 0.25 mg.; Drug: Recombinant choriogonadotropin alfa; Drug: Micronized natural progesterone.
- hMG ,Ganirelix,choriogonadotropin alfa,progesterone (Active Comparator): Human Menopausal Gonadotropin (hMG). Dose: 300 IU/24h from the 2nd day of the cycle throughout the stimulation.
  Ganirelix 0.25 mg,Dose: 250μg/24h since the day observe a follicle> 14mm. Recombinant choriogonadotropin alfa,Dose: 6,500 IU, pods, when follicles> 17 mm are observed.
  Micronized natural progesterone. Route of administration: vaginal. Dose: 400mg/24, from embryo transfer until the day of b-hCG.
  Interventions: Drug: Ganirelix 0.25 mg.; Drug: Recombinant choriogonadotropin alfa; Drug: Micronized natural progesterone.

INTERVENTIONS:
Drug: Ganirelix 0.25 mg. — Ganirelix 0.25 mg. Route of administration: Subcutaneous use. Dose: 250μg/24h since the day observe a follicle> 14mm.
  Other Names: ORGALUTRAN®.
Drug: Recombinant choriogonadotropin alfa — Recombinant choriogonadotropin alfa. Route of administration: Subcutaneous use. Dose: 6,500 IU, pods, when follicles> 17 mm are observed
  Other Names: OVITRELLE®.
Drug: Micronized natural progesterone. — Micronized natural progesterone. Route of administration: vaginal . Dose: 400mg/24, from embryo transfer until the day of b-hCG.
  Other Names: PROGEFFIK®.

SUMMARY:
Patients who have had or are expected to have a poor ovarian response (POR), because they meet any of the criteria of Bologna, can benefit from ovarian stimulation with 150 mg of alpha Corifollitropin (CFA) (Elonva ®) as single dose for a week, in the cycles of in vitro fertilization (IVF).

In this study aims to demonstrate non-inferiority of the Corifollitropin Alpha (CFA ) versus daily administration of Human Menopausal Gonadotropin (hMG) (Menopur ®) during the first seven days of ovarian stimulation, in a protocol with gonadotropin-releasing hormone ( GnRH) antagonists

DETAILED DESCRIPTION:
One of the most significant problems in fertilization treatments is Controlled Ovarian Stimulation low responsiveness . The incidence of low ovarian response is estimated at around 10-25%.The wide range of prevalence reported in the literature can be explained by the lack of consensus existed as to the criteria for the low response.

The ovarian response to gonadotropin stimulation is crucial for successful assisted reproduction techniques .Cycles with low rates response was obtained and increased cancellation rate and worst pregnancy rates .

Different criteria for the definition of low response, different tests to assess ovarian reserve and different threshold values for each has been used.

In 2010 a group of experts from the ESHRE ,achieved consensus on the criteria for low ovarian response to homogenize the study groups and reach meaningful conclusions, are known as "The Bologna criteria" ,they defined the "Poor Ovarian Response" (POR).

There is not sufficient to recommend most of the proposed treatments to improve pregnancy rates in poor responders evidence.

Taking into account the profile of equivalence and safety of CFA (Corifollitropin Alpha , active of ELONVA ® ) , different studies had been concluded that CFA can be an alternative to daily injections of recombinant follicle stimulating hormone ( rFSH) in normal responders patients in vitro fertilization cycle with ovarian stimulation.But more research is needed to determine whether long-acting recombinant follicle stimulating hormone ( rFSH) is safe and effective for use in women with low and high response.

The ovarian controlled stimulation with Alpha Corifollitropin produces significantly more oocytes compared to recombinant follicle stimulating hormone (r FSH ) administrated daily in normal responders patients, For this reason , the use of Alpha Corifollitropin may be beneficial in patients with poor response which the number of oocytes retrieved is crucial for successful treatment

There have been two studies in which the results are compared after ovarian stimulation with daily rFSH vs CFA . In both shows , retrospectively and prospectively , the CFA seems to be at least as effective as hMG recombinant follicle stimulating hormone ( rFSH) daily.

There are scientific publications showing that the association of luteinizing hormone ( LH) to recombinant follicle stimulating hormone ( rFSH) can improve embryos quality and achieved better pregnancy rate . The pregnancy rate was not statistically significant , in normal responders patients.

Recently reported the beneficial effect in POR patients treated with CFA and hMG.

The IVF treatment is known to affects the physical and mental condition in patients with infertility , being the excess emotional stress one of the most important reasons for discontinuation of treatment.

The ovarian stimulation with CFA simplifies treatment , reducing the administration of multiple daily injections ,and may reduce the emotional burden on patients.

ELIGIBILITY:
Inclusion Criteria:

1. - Age ≥ 18 years old.
2. - Signed informed consent to perform IVF and participation in this study.
3. - Due to characteristics of our center not perform treatments in patients

   * 40 years old ,and being one of the Bologna criteria that we will not be able to consider ,we decided to include patients affected subsidiary infertility treatment by IVF or intracytoplasmatic sperm injection (ICSI), present one of the following factors

     1. Have a history of surgical or medical treatment as a risk factor for POR.
     2. Patients witch had have a poor ovarian response in response to the ovarian controlled stimulation (previous cycle after conventional stimulation with ≤ 3 oocytes)
     3. Patients with ovarian reserve test anti-mullerian hormone(AMH ) <1.1 ng / ml (<8 pM) or antral follicle count (AFC)<7

Exclusion Criteria:

1. -Anovulation.
2. -Patient with tubal factor, untreated
3. -Patient with uterine pathology untreated
4. - Couples with severe male factor, fresh count <5 million / ml, and azoospermia in which the patient's sperm, epididymal or testicular is used

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of evolutionary gestation in each cycle | 20 week of gestation
  Evolutionary pregnancy has been defined as gestation of at least 1 fetus reaches 20 weeks of gestation diagnosed by normal ultrasound or confirmed by live birth
oocytes (MII) rate by patient | participants will be followed for the duration of the cycle,an expected average of 8-16 days.
  When follicular puncture occurs, we value the number of punctured follicles, total oocytes and MII oocytes

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | participants will be followed for the duration of the cycle,an expected average of 16 days.

CONTACTS AND LOCATIONS:
Overall Officials: Roser Taroncher, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Human Reproduction Unit of the La Fe University and Politechnic Hospital, Valencia, Spain

REFERENCES:
- [Background] Cousineau TM, Domar AD. Psychological impact of infertility. Best Pract Res Clin Obstet Gynaecol. 2007 Apr;21(2):293-308. doi: 10.1016/j.bpobgyn.2006.12.003. Epub 2007 Jan 22. PMID 17241818
- [Background] Devroey P, Boostanfar R, Koper NP, Mannaerts BM, Ijzerman-Boon PC, Fauser BC; ENGAGE Investigators. A double-blind, non-inferiority RCT comparing corifollitropin alfa and recombinant FSH during the first seven days of ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2009 Dec;24(12):3063-72. doi: 10.1093/humrep/dep291. Epub 2009 Aug 14. PMID 19684043
- [Background] Devroey P, Fauser BC, Platteau P, Beckers NG, Dhont M, Mannaerts BM. Induction of multiple follicular development by a single dose of long-acting recombinant follicle-Stimulating hormone (FSH-CTP, corifollitropin alfa) for controlled ovarian stimulation before in vitro fertilization. J Clin Endocrinol Metab. 2004 May;89(5):2062-70. doi: 10.1210/jc.2003-031766. PMID 15126522
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Keay SD, Liversedge NH, Mathur RS, Jenkins JM. Assisted conception following poor ovarian response to gonadotrophin stimulation. Br J Obstet Gynaecol. 1997 May;104(5):521-7. doi: 10.1111/j.1471-0528.1997.tb11525.x. No abstract available. PMID 9166190
- [Background] Kim CH, Jeon GH, Cheon YP, Jeon I, Kim SH, Chae HD, Kang BM. Comparison of GnRH antagonist protocol with or without oral contraceptive pill pretreatment and GnRH agonist low-dose long protocol in low responders undergoing IVF/intracytoplasmic sperm injection. Fertil Steril. 2009 Nov;92(5):1758-60. doi: 10.1016/j.fertnstert.2009.05.013. Epub 2009 Jun 12. PMID 19523618
- [Background] Kolibianakis EM, Venetis CA, Bosdou JK, Zepiridis L, Chatzimeletiou K, Makedos A, Masouridou S, Triantafillidis S, Mitsoli A, Tarlatzis BC. Corifollitropin alfa compared with follitropin beta in poor responders undergoing ICSI: a randomized controlled trial. Hum Reprod. 2015 Feb;30(2):432-40. doi: 10.1093/humrep/deu301. Epub 2014 Dec 9. PMID 25492411
- [Background] Kyrou D, Kolibianakis EM, Venetis CA, Papanikolaou EG, Bontis J, Tarlatzis BC. How to improve the probability of pregnancy in poor responders undergoing in vitro fertilization: a systematic review and meta-analysis. Fertil Steril. 2009 Mar;91(3):749-66. doi: 10.1016/j.fertnstert.2007.12.077. Epub 2008 Jul 21. PMID 18639875
- [Background] Mahmoud Youssef MA, van Wely M, Aboulfoutouh I, El-Khyat W, van der Veen F, Al-Inany H. Is there a place for corifollitropin alfa in IVF/ICSI cycles? A systematic review and meta-analysis. Fertil Steril. 2012 Apr;97(4):876-85. doi: 10.1016/j.fertnstert.2012.01.092. Epub 2012 Jan 23. PMID 22277766
- [Background] Pandian Z, McTavish AR, Aucott L, Hamilton MP, Bhattacharya S. Interventions for 'poor responders' to controlled ovarian hyper stimulation (COH) in in-vitro fertilisation (IVF). Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004379. doi: 10.1002/14651858.CD004379.pub3. PMID 20091563
- [Background] Pellicer A, Lightman A, Diamond MP, Russell JB, DeCherney AH. Outcome of in vitro fertilization in women with low response to ovarian stimulation. Fertil Steril. 1987 May;47(5):812-5. doi: 10.1016/s0015-0282(16)59170-5. PMID 3106105
- [Background] Pellicer A, Ardiles G, Neuspiller F, Remohi J, Simon C, Bonilla-Musoles F. Evaluation of the ovarian reserve in young low responders with normal basal levels of follicle-stimulating hormone using three-dimensional ultrasonography. Fertil Steril. 1998 Oct;70(4):671-5. doi: 10.1016/s0015-0282(98)00268-4. PMID 9797096
- [Background] Polyzos NP, De Vos M, Corona R, Vloeberghs V, Ortega-Hrepich C, Stoop D, Tournaye H. Addition of highly purified HMG after corifollitropin alfa in antagonist-treated poor ovarian responders: a pilot study. Hum Reprod. 2013 May;28(5):1254-60. doi: 10.1093/humrep/det045. Epub 2013 Feb 26. PMID 23442756
- [Background] Polyzos NP, Devos M, Humaidan P, Stoop D, Ortega-Hrepich C, Devroey P, Tournaye H. Corifollitropin alfa followed by rFSH in a GnRH antagonist protocol for poor ovarian responder patients: an observational pilot study. Fertil Steril. 2013 Feb;99(2):422-6. doi: 10.1016/j.fertnstert.2012.09.043. Epub 2012 Oct 16. PMID 23084565
- [Background] Pouwer AW, Farquhar C, Kremer JA. Long-acting FSH versus daily FSH for women undergoing assisted reproduction. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD009577. doi: 10.1002/14651858.CD009577.pub2. PMID 22696386
- [Background] Requena A, Landeras JL, Martinez-Navarro L, Calatayud C, Sanchez F, Maldonado V, Munoz M, Fernandez M, Gonzalez A, Lopez S, Lopez R, Pacheco A, Calderon G, Martinez V. Could the addition of hp-hMG and GnRH antagonists modulate the response in IVF-ICSI cycles? Hum Fertil (Camb). 2010 Mar;13(1):41-9. doi: 10.3109/14647270903586356. PMID 20384441
- [Background] Tarlatzis BC, Zepiridis L, Grimbizis G, Bontis J. Clinical management of low ovarian response to stimulation for IVF: a systematic review. Hum Reprod Update. 2003 Jan-Feb;9(1):61-76. doi: 10.1093/humupd/dmg007. PMID 12638782